CLINICAL TRIAL: NCT05000203
Title: Randomized Controlled Trial Comparing a Specific Intervention by Midwife to Address the Fear of Childbirth.
Brief Title: Intervention by Midwife to Address the Fear of Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Las Palmas de Gran Canaria (Other)
Collaborators: Servicio Canario de Salud (Other)
Responsible Party: Principal Investigator, Sergio Mies Padilla, Principal Investigator, University of Las Palmas de Gran Canaria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Código CEIm HUGCDN: 2021-169-1
Record Dates: First submitted 2021-07-08; First posted 2021-08-11 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Fear of Childbirth
Keywords: Fear; Childbirth; Midwifery; Education; Support

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A single blind will be performed by masking the data analysis. It will not be carried out in blinding of the participants due to impossibility given the nature of the education study. As far as possible, the control group will not be identified as pregnant women with severe fear of childbirth in the delivery area, since it is about receiving the usual care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific intervention for fear of childbirth (Experimental): Online education intervention Participants randomly assigned to the experimental group will be informed by telephone call of their inclusion in the first phase of the trial.
  Participants in the intervention group will be encouraged to attend routine consultations with their midwife and obstetrician, as well as to take advantage of the group maternal education that participants usually develop in their health center.
  Specific intranatal support
  An experimental group will be carried out with a specific support intervention in the obstetric-gynecological emergency area that will supplement the one usually provided to all pregnant women.
  At the end of the participant's stay within the emergency area due to hospital discharge, admission to the ward, or the end of the pregnancy, the collaborating midwife will fill out an online form designed to monitor the care offered. Said form will also be completed at the end of the work shift if the participant's care continues.
  Interventions: Behavioral: Online prenatal specific education; Behavioral: Intrapartum specific support
- Routine intervention for fear of childbirth (Active Comparator): Usual care
  Participants randomly assigned to the control group will be informed by telephone call of their inclusion in the first phase of the trial. The process under study will be explained in detail, resolving any doubts at that time.
  Regular intranatal support
  The participants in the control group will not be identified as pregnant women with fear of childbirth, and will receive the usual care in the obstetric-gynecological emergency area.
  Interventions: Behavioral: Prenatal usual education; Behavioral: Intrapartum usual support

INTERVENTIONS:
Behavioral: Online prenatal specific education — The sessions will start around 30 weeks of gestation with the intention that around 35-37 weeks all pregnant women have had the opportunity to attend all the sessions.
  Five specific online group sessions have been established for the fear of childbirth, each divided into three parts, and lasting approximately 60 minutes. In the first part, the aspects that are most relevant according to the reported experience of women with fear of childbirth will be discuss. In a second part, videos will be displayed starring midwives who will collaborate in specific intrapartum support with the aim of presenting the personnel involved in the care of women during delivery and immediate postpartum, and where the procedures and options available in the obstetric service of HUMIC. The session will end with brief therapy tasks. After each session, written documentation on the topics discussed will be made available to the participants.
  Arms: Specific intervention for fear of childbirth
Behavioral: Intrapartum specific support — At first, a group of expert midwives will be formed in support of pregnant women with fear of childbirth. The objective is that three midwives from each work group shift will include the women from the experimental group in the intrapartum support team. The working group will receive a seminar given by the researcher where the study protocol and an update on fear of childbirth will be explained, which will include information on: concept and prevalence, risk factors, consequences, diagnosis and treatment.
  For the follow-up of the participants, an instant messaging group will be formed where the collaborating midwives and the main researcher will be able to find out the existence of a participant within the emergency area or in the maternity ward, facilitating continued care in the changes of guard
  Arms: Specific intervention for fear of childbirth
Behavioral: Prenatal usual education — The participants in this group will follow the development of the usual interventions by midwives and obstetricians according to the established protocol for monitoring the pregnancy and / or by the private care system, as well as additional consultations for complications in pregnancy or consultations on demand that are considered necessary Group maternal education is offered in primary care center starting at week 28 of gestation. Although its content is supported by the Affective-Sexual and Reproductive Health Care Program, midwives are responsible for preparing the sessions according to their criteria to adapt them to the population. In addition to group interventions, pregnant women in the intervention environment also receive individualized educational attention in follow-up and control visits. After delivery, an inquiry will be made about the maternal education received by pregnant women during their current pregnancy.
  Arms: Routine intervention for fear of childbirth
Behavioral: Intrapartum usual support — A routine detection of fear of childbirth or a protocolized practice for this problem is currently not contemplated in the trial setting. The different professionals who pay their attention to the pregnant woman can detect the fear of childbirth thanks to their experience or different indicators such as the expression of fears by the pregnant woman, being able to offer individualized attention and resources for the approach, according to their awareness of the problem .
  Arms: Routine intervention for fear of childbirth

SUMMARY:
The main objective of the research is to implement a specific intervention directed by midwives to address the fear of childbirth in the prenatal and intrapartum periods. The results obtained in the specific intervention group under study will be compared with those of the control group that will follow the usual care.

Fear of childbirth is defined as a state of intense anxiety that leads some women to fear childbirth, provoking a response that can influence the course of pregnancy, childbirth, and postpartum, as well as well-being and child development. Beneficial results have been shown in counseling, and prenatal education for childbirth, appropriate therapies to prevent, or at least reduce this suffering and its consequences. These interventions must be specific to see an improvement in symptoms, and must use a combination of various approaches to promote not only a reduction in fear, but a positive birth experience.

The population under study will be made up of pregnant women with a fear of childbirth detected in the second trimester of gestation. The sample will be recruited in the area of prenatal diagnosis of the Hospital Materno Infantil of Canarians (HUMIC). The start of the recruitment of participants is expected in June 2021, the online prenatal education intervention in August 2021 and the intrapartum intervention in October 2020. The intervention is expected to end in April 2022. It will be carried out a consecutive sampling until reaching the estimated sample size of 190 participants with fear of severe delivery who will be randomized to one of the two arms of the trial.

DETAILED DESCRIPTION:
A parallel group randomized controlled trial will be conducted in a cohort of women with a high level of fear of childbirth. Participants will be randomized to one of two arms: specific intervention group or usual care control group.

Initially, the fear of childbirth and associated factors will be evaluated in the second trimester of pregnancy, between weeks 20 and 24 of gestation. This will be followed by prenatal intervention in women who meet the inclusion criteria. In the intervention group, it will begin around week 30 of gestation, supplementing the interventions that are usually offered to all pregnant women, and that the control group will also receive. The results of the prenatal phase will be evaluated by means of the changes in the value of fear of childbirth in each group.

The intranatal intervention begins after 37 weeks of gestation, once the pregnant women attend the obstetric-gynecological emergency service. The participants will remain in the same group assigned in the first part, intervention or intrapartum control. The efficacy of the intervention will be evaluated after delivery by comparing the changes in the value of fear of childbirth, experience, satisfaction, and obstetric and neonatal outcomes between both groups.

Secondarily, an observational, descriptive study is proposed, with an analytical component and a cross section on aspects such as: the factors detected in the pregnant women who participated in the initial evaluation of fear of childbirth, the aspects related to the care received during pregnancy and childbirth in the participants of both groups, and the information obtained in the evaluation of the experience of midwives about fear of childbirth as well as the details of the intrapartum care offered during the study.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* 20-24 weeks of gestation
* Fear of childbirth
* Normal morphological ultrasound.

Exclusion Criteria:

* Online questionnaire disability
* Videoconference disability
* Incomplete questionnaires
* Language barrier.

Withdrawal criteria:

* Elective caesarean section
* Delivery before 37 weeks of gestation
* Non-attendance at educational sessions
* Delivery in a place other than HUMIC
* Fetal death
* Decline of informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Change in the value of fear of childbirth | At 20-24 and 37 weeks gestation
  Describe and compare the value of fear of childbirth measured by the Wijma Expectations Questionnaire in version A in its validated version into Spanish, in the prenatal education intervention group and in the control group between 20-24 weeks of gestation and 37 weeks of gestation. The questionnaire is made up of 31 questions and establishes values from 0 to indicate a lower fear of childbirth to 155, which indicates the maximum value of fear of childbirth.
Value of fear of postnatal childbirth | Before 10 days postpartum
  Describe and compare the value of fear of postnatal childbirth measured by the Wijma Experience Questionnaire in version B, in its validated version into Spanish, in the intranatal intervention group and in the control group.The questionnaire is made up of 33 questions and establishes values from 0 to indicate a lower fear of childbirth to 165, which indicates the maximum value of fear of childbirth.
Postpartum maternal satisfaction | Before 10 days postpartum
  Evaluate and Compare maternal satisfaction in both study groups using Childbirth Experience Questionnaire in its validated version into Spanish. Satisfaction is evaluated through 22 questions, the highest score of 88 reporting greater satisfaction, and the lowest score of 22 reporting less satisfaction.
Obstetric outcomes of childbirth | Before 10 days postpartum
  Describe and compare the following obstetric outcomes of childbirth between both study groups: type of onset of delivery, epidural use, use of oxytocin, type of completion of delivery, gestational giving to delivery, perineal tear, episiotomy, total duration of delivery
Neonatal outcomes of childbirth | Before 10 days postpartum
  Describe and compare the following neonatal outcomes of childbirth between both study groups

SECONDARY OUTCOMES:
Description of the sociodemographic data of the participants in the recruitment for the trial.. | At 20-24 weeks gestation
  Description of sociodemographic data of the participants in the sample collection for the trial. The data of all women who fill out the online form in the second trimester of pregnancy will be included.
Description of obstetrics data of the participants in the recruitment for the trial. | At 20-24 weeks gestation
  Description of obstetrics data of the participants in the sample collection for the trial. The data of all women who fill out the online form in the second trimester of pregnancy will be included. It includes the assessment of parity, and the type of completion of their last birth in case of multiparous women
Description of the birthing preferences of the participants in the recruitment for the trial. | At 20-24 weeks gestation
  Description of birthing preferences of the participants in the sample collection for the trial. The data of all women who fill out the online form in the second trimester of pregnancy will be included. The preferred mode of delivery will be evaluated by the question with four answer options: vaginal delivery, probably vaginal delivery, probably cesarean delivery, or cesarean delivery. Thinking about place to give birth will be evaluated with response options: public hospital, private clinic, or home.
Description of the previous birth experiences of the participants in the recruitment for the trial. | At 20-24 weeks gestation
  Description of the previous birth experiences of the participants in the sample collection for the trial. The data of all women who fill out the online form in the second trimester of pregnancy will be included. The previous birthing experience it will be evaluated by the linear scale from 1 (very negative) to 5 (very positive). The satisfaction in previous delivery will be evaluated by choosing a value on a linear scale ranging from 1 (very dissatisfied) to 5 (very satisfied).
Compare the change in value of fear of part before and after delivery. | Before 10 days postpartum
  Compare the results of measuring fear of childbirth before and after childbirth between the study groups.The value of fear before childbirth will be measured by the Wijma Expectations Questionnaire in version A in its validated version into Spanish, in the prenatal education intervention group and in the control group in 37 weeks of gestation obtained in outcome measure 1. The value of fear after childbirth will be measured by the Wijma Experience Questionnaire in version B in its validated version into Spanish in the intranatal intervention group and in the control group obtained in outcome measure 2. To compare both measurements, the scores obtained will be normalized
Intrapartum intervention performed by midwives | During the intrapartum intervention, an average of 6 months
  To describe the intrapartum interventions performed by the midwives during the individual care of each pregnant woman in the intervention group. After each support the midwives will fill out a form with the following questions: identify the name of the midwife, day, work shift, time that the collaborating midwife contacts the participant, reason for consultation, and procedures performed during their care to reduce the fear of childbirth.

OTHER OUTCOMES:
Prenatal education received childbirth. | At 37 weeks gestation
  To evaluate prenatal education received in both study groups. Questions about her attendance at regular maternal education classes, the topics discussed in her or with the midwife individually, and the advice received to improve coping with her fear of childbirth.
Experience of the midwives before the start of the intervention | For 30 days
  To evaluate the experience in the care of women with fear of childbirth of midwives who provide care in the area of delivery by adapting a questionnaire based on a study that investigates the practices and knowledge of midwives in relation to the subject matter (d Vries, 2020)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Mies Padilla, Matrona, Principal Investigator — Matrona asistencial del área del paritorio del Hospital Materno Infantil de Gran Canaria
Locations (1):
- Hospital Materno Infantil de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: Yes
It is planned to share the training plan of the online sessions
Supporting Information: Study Protocol
Time Frame: After publication of results
Access Criteria: Health professionals

REFERENCES:
- [Result] Mies Padilla S, Gonzalez de la Torre H, Lopez Alcaide E, Verdu Soriano J, Martin Martinez A. Randomized Controlled Trial of Interventions Used by Midwives to Treat Fear of Childbirth. Nurs Res. 2024 Nov-Dec 01;73(6):E221-E231. doi: 10.1097/NNR.0000000000000756. Epub 2024 Jul 17. PMID 39103313